CLINICAL TRIAL: NCT06584123
Title: Exploring the Potential for 18F-fluoro-ethyl-tyrosine (18F-FET) to Enable Wider Access to Molecular Imaging for Patients With Pituitary Adenomas (FET-pit-PET Study)
Brief Title: Molecular Pituitary Imaging Using 18F-FET PET
Acronym: FET-pit-PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Mark Gurnell, Professor of Clinical Endocrinology, University of Cambridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24/LO/0542
Record Dates: First submitted 2024-07-24; First posted 2024-09-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pituitary Adenoma
Keywords: Molecular pituitary imaging; Functional pituitary imaging; 18F-FET PET
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient's who have previously undergone 11C-Methionine PET during routine clinical care will be invited to undergo 18F-Fluoro-ethyl-tyrosine PET (FET PET).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study cohort (Experimental): All patient's enrolled in the study will undergo an 18F-FET-PET
  Interventions: Diagnostic Test: 18F-Fluoro-ethyl-tyrosine (FET) PET

INTERVENTIONS:
Diagnostic Test: 18F-Fluoro-ethyl-tyrosine (FET) PET — 18F-Fluoro-ethyl-tyrosine PET study of the pituitary

SUMMARY:
The goal of this single centre pilot study is to explore whether 18F-fluoro-ethyl-tyrosine PET (FET-PET) yields comparable findings to 11C-methionine PET (Met-PET) for the localisation of pituitary tumours.

DETAILED DESCRIPTION:
Up to 20 patients with pituitary adenomas (PA) who have previously undergone 11C-methionine PET (Met-PET) as part of routine clinical care will undergo 18F-fluoroethyltyrosine PET (FET-PET). Patients with newly diagnosed PA or residual/recurrent pituitary tumours following previous treatment will be eligible for recruitment to the study.

Quantitative and qualitative analyses will be performed to assess whether MET-PET and FET-PET yield comparable findings in patients with newly diagnosed or recurrent PA.

ELIGIBILITY:
Inclusion criteria

* Participant is willing and able to give informed consent for participation in the study
* Male or female, age 18 or above
* Presence of pituitary adenoma suspected on the basis of clinical/biochemical and/or radiological findings
* Previous 11C-Met-PET/CT

Exclusion criteria

* Inability to give informed consent
* Pregnancy or suspected pregnancy
* Inability to lie supine for 30-60 minutes
* Patient body habitus above scanner dimensions
* Known allergy to intravenous radiographic contrast agents

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Standardized Uptake Values (SUVmax) over pituitary tumour on each of 11C-methionine and 18F-fluoroethyltyrosine PET scans | 1 day
  Comparison of maximum Standardized Uptake Values (SUVmax) measured over pituitary tumours on each type of PET scan.

SECONDARY OUTCOMES:
Maximum Standardized Uptake Values (SUVmax) over normal pituitary gland and parasellar structures (e.g. cavernous sinuses) on each of 11C-methionine and 18F-fluoroethyltyrosine PET scans | 1 day
  Comparison of maximum Standardized Uptake Values (SUVmax) measured over normal pituitary gland and parasellar structures (e.g. cavernous sinuses) on each type of PET scan.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gurnell, MD, PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacFarlane J, Bashari WA, Senanayake R, Gillett D, van der Meulen M, Powlson AS, Kolias A, Koulouri O, Gurnell M. Advances in the Imaging of Pituitary Tumors. Endocrinol Metab Clin North Am. 2020 Sep;49(3):357-373. doi: 10.1016/j.ecl.2020.06.002. Epub 2020 Jul 15. PMID 32741476
- [Background] Koulouri O, Kandasamy N, Hoole AC, Gillett D, Heard S, Powlson AS, O'Donovan DG, Annamalai AK, Simpson HL, Akker SA, Aylwin SJ, Brooke A, Buch H, Levy MJ, Martin N, Morris D, Parkinson C, Tysome JR, Santarius T, Donnelly N, Buscombe J, Boros I, Smith R, Aigbirhio F, Antoun NM, Burnet NG, Cheow H, Mannion RJ, Pickard JD, Gurnell M. Successful treatment of residual pituitary adenoma in persistent acromegaly following localisation by 11C-methionine PET co-registered with MRI. Eur J Endocrinol. 2016 Nov;175(5):485-498. doi: 10.1530/EJE-16-0639. Epub 2016 Aug 25. PMID 27562400
- [Background] Koulouri O, Steuwe A, Gillett D, Hoole AC, Powlson AS, Donnelly NA, Burnet NG, Antoun NM, Cheow H, Mannion RJ, Pickard JD, Gurnell M. A role for 11C-methionine PET imaging in ACTH-dependent Cushing's syndrome. Eur J Endocrinol. 2015 Oct;173(4):M107-20. doi: 10.1530/EJE-15-0616. Epub 2015 Aug 5. PMID 26245763
- [Background] Koulouri O, Hoole AC, English P, Allinson K, Antoun N, Cheow H, Burnet NG, Donnelly N, Mannion RJ, Gurnell M. Localisation of an occult thyrotropinoma with 11C-methionine PET-CT before and after somatostatin analogue therapy. Lancet Diabetes Endocrinol. 2016 Dec;4(12):1050. doi: 10.1016/S2213-8587(16)30311-4. Epub 2016 Oct 21. No abstract available. PMID 27777050
- [Background] Bashari WA, Senanayake R, Koulouri O, Gillett D, MacFarlane J, Powlson AS, Fernandez-Pombo A, Bano G, Martin AJ, Scoffings D, Cheow H, Mendichovszky I, Tysome J, Donnelly N, Santarius T, Kolias A, Mannion R, Gurnell M. PET-guided repeat transsphenoidal surgery for previously deemed unresectable lateral disease in acromegaly. Neurosurg Focus. 2020 Jun;48(6):E8. doi: 10.3171/2020.3.FOCUS2052. PMID 32480379
- [Background] Grosu AL, Astner ST, Riedel E, Nieder C, Wiedenmann N, Heinemann F, Schwaiger M, Molls M, Wester HJ, Weber WA. An interindividual comparison of O-(2-[18F]fluoroethyl)-L-tyrosine (FET)- and L-[methyl-11C]methionine (MET)-PET in patients with brain gliomas and metastases. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1049-58. doi: 10.1016/j.ijrobp.2010.07.002. Epub 2011 May 11. PMID 21570201
- [Background] Currie GM, Trifunovic M, Kiat H, Saunders C, Chung D, Ong YY, Wilkinson M, Witte K, Magnussen J. Pituitary incidentaloma found on O-(2-18F-fluoroethyl)-l-tyrosine PET. J Nucl Med Technol. 2014 Sep;42(3):218-22. doi: 10.2967/jnmt.113.136291. Epub 2014 Jun 19. PMID 24948822
- [Background] van den Bergh AC, Pruim J, Links TP, van der Vliet AM, Sluiter W, Wolffenbuttel BH, Langendijk JA, Hoving EW, Dullaart RP. Tyrosine positron emission tomography and protein synthesis rate in pituitary adenoma: different effects of surgery and radiation therapy. Radiother Oncol. 2011 Feb;98(2):213-6. doi: 10.1016/j.radonc.2010.12.020. Epub 2011 Feb 4. PMID 21296442